CLINICAL TRIAL: NCT07006155
Title: Intra-individual Comparison of PET Scans on the Biograph Vision 600 With the New Biograph Vision.X PET/CT
Brief Title: Biograph Vision 600 Versus Biograph Vision.X PET/CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valentina Garibotto (Other)
Responsible Party: Sponsor-Investigator, Valentina Garibotto, Director of the Division of Nuclear Medicine and Molecular imaging, associate professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-D00005
Record Dates: First submitted 2025-04-07; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Alzheimer Disease
Keywords: PET/CT; Vision; image quality; diagnostic performance
MeSH Terms: conditions — Neoplasms; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vision X (Experimental): PET/CT images acquired with Vision.X
  Interventions: Device: Images
- Vision 600 (Active Comparator): PET/CT images in Vision 600
  Interventions: Device: Images

INTERVENTIONS:
Device: Images — PET/CT images

SUMMARY:
The main purpose is to evaluate initial clinical experiences and to explore whether the Vision.X system yields improved image quality and diagnostic performance compared to Vision 600.

ELIGIBILITY:
Inclusion Criteria:

* Written Inform Consent to participating.
* 18 to 85 years of age
* Willing and able to comply with the requirements of the study, as judged by the investigator

Exclusion Criteria:

* Women in pregnancy
* Patients unable to lie still for the duration of the examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
change of physician's diagnostic confidence | through study completion , an average of 1 year
  The primary outcome will be image quality assessed on the two compared PET systems, namely Vision and Vision X.
  For the all PET scans, three independent, blinded physicians will evaluate the scans and establish diagnoses. They will assess the following quality criteria using 5-point Likert scales:
  * Overall Image Quality: 1 = poor, 5 = excellent,
  * Image Noise: 1 = excessive noise, 5 = no perceptible noise, Image quality is associated with physician's diagnostic confidence and with the ability to detect smaller lesions that can lead to more accurate staging of diseases, particularly in oncology and neurology. This enhanced staging can influence treatment decisions, allowing healthcare professionals to tailor interventions based on a more precise understanding of the extent and location of the disease.

SECONDARY OUTCOMES:
lowering of the radiotracer activity | through study completion , an average of 1 year
  The secondary outcome will be the assessment of image quality (as for the primary outcome) on simulated lower doses of radiotracer activity on both PET systems (Vision and Vision X).
  To assess this, the same parameters described in section 5.1 will be evaluated across different emulated scan times, as shorter scanning times allow simulating lower administered activities. These will be generated by binning the list-mode data with varying frame durations for both scanner acquisitions.
  The lowering of the radiotracer activity maintaining a high-quality image is relevant for its capacity to reduce the radiation exposure for the patients and contributes to optimizing healthcare resources.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided